CLINICAL TRIAL: NCT01225653
Title: Topical Application of Latanoprost in Diabetic Retinopathy
Acronym: Latano-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Latano-2; 2010-022433-29 (EudraCT Number)
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Diabetic Retinopathy
Keywords: Latanoprost; vasodilation; diabetic retinopathy
MeSH Terms: conditions — Diabetic Retinopathy; Aneurysm | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Latanoprost (Experimental): Topical treatment with latanoprost
  Interventions: Drug: Latanoprost
- Placebo (Placebo Comparator): Placebo arm
  Interventions: Drug: Latanoprost

INTERVENTIONS:
Drug: Latanoprost — Topical application
  Other Names: No other names

SUMMARY:
Randomized double-blinded two-year intervention study with topical application of latanoprost or placebo eye drops in patients with diabetic retinopathy.

DETAILED DESCRIPTION:
The primary objective is to study if a sustained contraction of pathologically dilated retinal arterioles can be obtained. Retinal arteriolar diameter and the diameter response to increased blood pressure is studied using the Dynamic Vessel Analyzer (Imedos, Germany.

The secondary objective is to study whether the intervention can halt the development of diabetic retinopathy, which is assessed by optical coherence tomography (OCT) scanning and fundus photography.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-36 years old
* Diabetes mellitus with retinopathy

Exclusion Criteria:

* Pregnancy
* Previous ocular disease other than diabetic retinopathy
* General disease with possible influence on the eye

Ages: 20 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2010-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The diameter of retinal arterioles | 24 months
  The diameter of retinal arterioles will be assessed using the Dynamic Vessel Analyzer

SECONDARY OUTCOMES:
The severity of diabetic retinopathy | 24 months
  Severity of diabetic retinopathy will be measured by optical coherence tomography (OCT) scanning and fundus photography

CONTACTS AND LOCATIONS:
Overall Officials: Toke Bek, Professor, Principal Investigator — Dept of Ophthalmology, Århus University Hospital
Locations (1):
- Department of Ophthalmology, Århus University Hospital, Aarhus, Denmark